CLINICAL TRIAL: NCT02275182
Title: Impact of Dexmedetomidine Sedation on the Post-Operative Cognition Dysfunction--a Multiple Center,Randomized, Controlled,Double Blinded Clinical Trial.
Brief Title: Impact of Dexmedetomidine on the Post-Operative Cognition Dysfunction(POCD) in Geriatric Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: The First Affiliated Hospital of Anhui Medical University (Other)
Responsible Party: Principal Investigator, Xinqi Cheng, Anesthesia Department, The First Affiliated Hospital of Anhui Medical University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 201401
Record Dates: First submitted 2014-10-21; First posted 2014-10-27 (Estimated); Last update posted 2018-04-25 (Actual); Status verified 2018-04

CONDITIONS: Postoperative Confusion; Delirium
Keywords: Dexmedetomidine
MeSH Terms: conditions — Delirium | interventions — Dexmedetomidine; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Dexmedetomidine (Experimental): 0.5μg/kg Dexmedetomidine as initial loading dose is given for 15 minutes before induction of anesthesia, followed by a maintenance infusion of 0.4μg/kg/h and stopped 30 minutes before the surgery over.
  Interventions: Drug: Dexmedetomidine
- Controlled (Placebo Comparator): 0.5μg/kg Saline as initial loading dose is given for 15 minutes before induction of anesthesia, followed by a maintenance infusion of 0.4μg/kg/h and stopped 30 minutes before the surgery over.
  Interventions: Drug: Saline

INTERVENTIONS:
Drug: Dexmedetomidine — 0.5μg/kg Dexmedetomidine as initial loading dose is given for 15 minutes before induction of anesthesia, followed by a maintenance infusion of 0.4μg/kg/min and stopped 30 minutes before the surgery over.
  Other Names: Yisi
  Arms: Dexmedetomidine
Drug: Saline — 0.5μg/kg saline as initial loading dose is given for 15 minutes before induction of anesthesia, followed by a maintenance infusion of 0.4μg/kg/min and stopped 30 minutes before the surgery over.
  Arms: Controlled

SUMMARY:
Post-Operative Cognition Dysfunction (POCD) is a common complication after surgery, POCD can lead to a reduced ability and seriously affect the quality of life of patients, increase personal and social burden, POCD may also increase mortality.POCD can occur at any age, but the long-term, affect the daily lives of POCD in elderly patients over 60 years of age are more prone. Age is a risk factor for advanced or long-term POCD. POCD determined by preoperative cognitive function and psychological scales postoperative assessment, the main recommendation of the agreed test methods include, Rey auditory verbal test, the connection test, digit span test. In this study, preoperative mini-mental state examination (MMSE) screening, comprehensive neurological function during hospitalization for memory, attention, executive function and exercise capacity test, and telephone follow-up after discharge Scale Revised (TICS-M) test.

Few study showed that dexmedetomidine may improve cognitive function in young patients others show that dexmedetomidine did not reduce POCD incidence after 24 hours of surgery. These results conflict and it is necessary to carry out large-scale, multi-center, randomized, controlled clinical study to determine whether dexmedetomidine reduce the POCD incidence or not for elderly patients.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent
2. Selective surgery and general anesthesia patients(abdomen,orthopedics and urology surgery is preferred）；
3. Age 65-90 yrs；
4. Anesthesia Society of American (ASA) Scale II~III；
5. Anticipated surgery time 2-6 hrs； -

Exclusion Criteria:

1. Dementia patients（Mini-mental state examination< 20）
2. Factors existed that affect cognition assessment such as language,visual,and auditory dysfunction；
3. Unstable metal status and mental disease；
4. The cognitive function examination in 3-6 months is not anticipated to be completed
5. II-III Atrioventricular block；
6. Heat rate < 50 beats/minutes；
7. Parkinson's Disease；
8. May occur or have occurred the difficult airway or anticipated delayed extubation
9. Sure or suspected abuse of analgesic and sedation drug；
10. Allergic to the trial drug and other anesthesia drug contraindication； -

Ages: 65 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 864 (Actual)
Dates: Start 2014-10 (Actual); Primary Completion 2017-01 (Actual); Study Completion 2017-02-20 (Actual)

PRIMARY OUTCOMES:
The change of incidence of postoperative cognition dysfunction | 1 day Before surgery,the 3rd,7th day after the surgery.
  1. The neuropsychological tests performed at the day before the surgery, the 3rd and 7th day after the surgery respectively.
  2. A test environment to keep quiet, well-lit, non-interference, all the test items should be completed within 30 min.
  3. Normal population (65 to 90 years age-matched 400 non-surgery people) should perform neuropsychological tests in the same time interval, then calculate the score difference(ΔXc), and the standard deviation(SD) of the difference.
  4. Calculate the difference(ΔX) between the score obtained before surgery and 3 or 7 days after the surgery (there are both positive and negative, we use the absolute value), with this difference( ΔX) divided by the standard deviation（SD）of the difference of the normal population, that is ΔX / SD and it is the Z score.
  5. POCD Diagnosis: if a patient has two or more than two of the absolute value of Z scores ≥1.96, the POCD is exist.
The change of incidence of postoperative delirium | The first, second and third day after the surgery.
  Through CAM-ICU to assess the incidence of the postoperative delirium.
The change of Neuropsychological status | the 3rd,6th month after the surgery
  Through the Telephone Interview for Cognitive Status-Modified(TICS-m) to follow up.

SECONDARY OUTCOMES:
The occurrence of cardiovascular events. | from begging of the anesthesia to the time the patients discharge, up to 1 month.
The incidence of any adverse or severe adverse events. | From the beginning of the admitted to 6 month after the surgery, up to 6 month.
  Including kidney or brain related adverse events.
The variation of heart rate. | From the beginning to the end of anesthesia,up to 6 hours.
  Heart rate is recorded every 15 minutes during the anesthesia.
The variation of blood pressure. | From the beginning to the end of anesthesia,up to 6 hours.
  blood pressure is recorded every 15 minutes during the anesthesia.
the variation of pulse oxygen saturation. | From the beginning to the end of anesthesia,up to 6 hours.
  Pulse oxygen saturation is recorded every 15 minutes during the anesthesia.
The monitor of depth of anesthesia. | From the beginning to the end of anesthesia,up to 6 hours.
  Bispectral index (Bis) is recorded every 15 minutes during the anesthesia.
The serum concentrations of BDNF | From the baseline to the 3-day,7-day and 1-month.
  Serum level of brain-derived neurotrophic factor (BDNF) was measured

CONTACTS AND LOCATIONS:
Overall Officials: Wei Er Gu, Principal Investigator — The First Affiliated Hospital of Anhui Medical University
Locations (13):
- China (13):
  - Anqing Municipal Hospital, Anqing, Anhui
  - Affiliated Hospital of Bengbu Medical College, Bengbu, Anhui
  - Affiliated Chaohu Hospital of Anhui Medical Hospital, Chaohu, Anhui
  - Binhu Hospital of Hefei, Hefei, Anhui
  - Second Affiliated Hospital of Anhui Medical University, Hefei, Anhui
  - The First Affiliated Hospital of Anhui Medical University, Hefei, Anhui
  - The first Hospital of Hefei, Hefei, Anhui
  - The Second Hospital of Hefei, Hefei, Anhui
  - The Second People's Hospital of Anhui, Hefei, Anhui
  - the people's Hospital of Liuan, Liuan, Anhui
  - the people's Hospital of Tongling, Tongling, Anhui
  - The First Affiliated Hospital of Wannan Medical College, Wuhu, Anhui
  - The second People's Hospital of Wuhu, Wuhu, Anhui